CLINICAL TRIAL: NCT00256841
Title: Dose Escalation of Xeloda or 5FU Continuous Infusion in Combination With Taxotere and Concurrent Once Weekly, Hypofractionated Chest Radiotherapy for Advanced Non Small Cell Lung Cancer: A Phase I/II Study
Brief Title: Hypo-Hyperfractionated Chest Radiation for Non Small Cell Lung Cancer With Taxotere/Xeloda Combination Chemotherapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Clinical Oncology Research Associates (Other)
Responsible Party: Principal Investigator, Paul Schwarzenberger, MD, Medical Oncologist, Clinical Oncology Research Associates
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hypo 2
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Hypofractionated Chest Radiation; Taxotere; 5-FU
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Radiotherapy

INTERVENTIONS:
Drug: Chemotherapy
Procedure: Radiation Therapy

SUMMARY:
The study is designed for patients with non small cell lung cancer whose cancer is too advanced and therefore cannot be operated with the goal of completely removing the cancer. At this stage of the disease, most patients cannot be cured from the disease, however, treatment can help to live longer and better by keeping the cancer under control. For that purpose, patients traditionally receive radiation therapy or chemotherapy or both treatments in succession. Recently, the administration of both treatment methods given concurrently showed somewhat better results when compared to successive administration. In some studies the drug Taxotere together with radiation performed well in keeping the cancer better under control.

Combination of the drug Taxotere together with a compound called 5-FU either as continuous infusion or in its oral form of a pill called "Xeloda" enhanced its anti cancer activity substantially.

One goal of this study is to investigate how much of the combination can be given in conjunction with chest radiation. Using X-rays, the study will also evaluate how much shrinkage of the cancer is caused by this treatment directly at the tumor site and other areas where the cancer may have also spread.

In this study the radiation will be given on only one day per week in two sessions, rather than divided over five days per week (Monday through Friday) as it is more commonly used. However, both schedules have been found to be equally effective.

The treatment program will use increasing doses of the 5-FU medication, either as infusion or as pill to find the highest dose that is tolerated. Once the highest tolerated dose is determined, subsequent patients who will be enrolled will continue to be treated at that dose level. The dose of the drug Taxotere will remain the same throughout.

Hypothesis: Our previous research suggests that the combination of Taxotere and 5-FU given together with weekly chest radiation will provide a more convenient form of treatment than the conventional approach and also be at least similar in its efficacy.

DETAILED DESCRIPTION:
The original once weekly hypofractionated chest irradiation protocol descrived by Salazar et al. will be followed with a slight modification. The dose will be split in two fractions, which will be given 6 hours apart. We found that this fractionation in two doses reduces radiation-related side effects. Treatment will be given to a large field with a 2-3 cm tumor margin. All involved or suspicious nodal areas will be radiated as well. A total of 12 treatments will be administered in weekly. Total treatment will be 6000 cGy. Radiation treatment will be administered within 2 hours of Taxotere infusion.

All patients will receive a fixed dose of Taxotere of 25 mg/m2 once per week on the day of radiotherapy preceeding the radiation. All patients will be premedicated using standard antiemetics and Decadron (8 mg po 12 hours prior Taxotere, 1 mg Kytril po, 20 mg Decadron iv , 50 mg Benadryl iv and 20 mg Pepcid iv , all 30 min prior Taxotere).

A dose escalation of 5-FU or Xeloda will be employed. 5-FU will be given as continuous infusion, Xeloda orally Monday through Friday throughout the 12 weeks of radiation. Upon reaching the maximum tolerated dose, the remainder of patients will be treated at the 5-FU/Xeloda dose level below the MTD.

Patients for who are unable to tolerate oral Xeloda because of the size of the tablets or difficulties with their upper gastroiontestinal tract or for whom Xeloda cannot be obtained, the intravenous equivalent of 5-Fluorouracil (5-FU) will be administered as a continuous intravenous infusion. Patients who started out on Xeloda and during the treatment experience difficulties in continuing taking Xeloda maybe switched to a biological equivalent dose of 5-FU during the treatment. The 5-FU dose range administered in lieu of Xeloda will be administered and adjustments will be made in 50 mg/m2/day steps as previously pubished by Lokich et al.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic evidence of NSCLC. Patients with bronchoalveolar type of NSCLCA are not eligible.
2. Should a second malignancy be present or discovered, subjects will only be eligible if the NSCLCA is determined by the PI to be the more life-threatening disease compared to the other malignancy in regards of life-expectancy.
3. All patients must have locally advanced disease (stage III A or III B) or metastatic (stage 4). Other stages are not eligible.
4. Performance status of 0 -1 (ECOG Criteria).
5. Patients should have an absolute granulocyte count > 1000/mm3 and a platelet count > 80,000/mm3.
6. Patients should have adequate hepatic function as indicated by a serum bilirubin < upper limit of normal (ULN); ALT and AST <2.5 ULN if alkaline phosphatase is < ULN. Alkaline phosphatase may be up to 4 x ULN if transaminases are < ULN. However, patients who have both transaminase elevation > 2 x ULN and alkaline phosphatase > 2.5 x ULN are not eligible for this study.
7. Subjects with with severe renal impairment (creatinine clearance below 30 mL/min [Cockroft and Gault]) are ineligible.
8. Patients should have at least a predicted FEV1 of 30%.
9. Patients with active ischemic heart disease (NYHA Class III or IV), congestive heart failure, symptomatic arrythmias, or a recent history of a myocardial infarction are excluded.
10. Patients with medically uncontrollable hypercoagalbility syndromes are not eligible. Patients who are on therapeutic anticoagulation are not excluded.
11. Patients with pre-existing serious adverse effects to 5-FU are not eligible for this study. Specifically, subjects with prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil.
12. Patients with medical contraindications to Taxanes are not eligible.
13. No other serious concurrent medical illness or active infection which would jeopardize the ability of the patient to receive with reasonable safety the chemotherapy and surgery program outlined in this protocol is allowed.
14. Subjects where studies or clinical examination demonstrates lack of physical integrity of the upper gastrointestinal tract, inability to swallow tablets or those who have malabsorption syndrome are not eligible.
15. Subjects who have had an organ allograft are not eligible.
16. Signed informed consent: each patient must be aware of the neoplastic nature of his/her disease and willingly consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
17. Pregnant women and nursing mothers are ineligible. Eligible patients of reproductive age should use contraception. Woman of childbearing potential with either a positive or no pregnancy test at baseline. Woman of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
18. Sexually active males unwilling to practice contraception during the study will not be eligible.
19. Patients must be at least 18 years old.
20. Known HIV positive patients will not be eligible.
21. Patients with prior treatment of Taxotere, Xeloda or 5FU will not be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Saftey

SECONDARY OUTCOMES:
Efficacy
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Paul Schwarzenberger, MD, Principal Investigator — CORA
Locations (1):
- Mobile Infirmary Medical Center, Mobile, Alabama, United States

REFERENCES:
- [Background] Schwarzenberger P, Theodossiou C, Barron S, Diethelm L, Boyle M, Harrison L, Wynn RB, Salazar OM, Fariss A. Dose escalation of docetaxel concomitant with hypofractionated, once weekly chest radiotherapy for non-small-cell lung cancer: a phase I study. Am J Clin Oncol. 2004 Aug;27(4):395-9. doi: 10.1097/01.coc.0000131943.02929.ac. PMID 15289734
- [Background] Salazar OM, Slawson RG, Poussin-Rosillo H, Amin PP, Sewchand W, Strohl RA. A prospective randomized trial comparing once-a-week vs daily radiation therapy for locally-advanced, non-metastatic, lung cancer: a preliminary report. Int J Radiat Oncol Biol Phys. 1986 May;12(5):779-87. doi: 10.1016/0360-3016(86)90036-2. PMID 3519551
- [Background] Salazar OM, Van Houtte P, Rubin P. Once-a-week radiation therapy for locally advanced lung cancer. Final report. Cancer. 1984 Aug 15;54(4):719-25. doi: 10.1002/1097-0142(1984)54:43.0.co;2-s. PMID 6744205
- [Background] Slawson RG, Salazar OM, Poussin-Rosillo H, Amin PP, Strohl R, Sewchand W. Once-a-week vs conventional daily radiation treatment for lung cancer: final report. Int J Radiat Oncol Biol Phys. 1988 Jul;15(1):61-8. doi: 10.1016/0360-3016(88)90347-1. PMID 2839442
- [Background] O'Shaughnessy J, Miles D, Vukelja S, Moiseyenko V, Ayoub JP, Cervantes G, Fumoleau P, Jones S, Lui WY, Mauriac L, Twelves C, Van Hazel G, Verma S, Leonard R. Superior survival with capecitabine plus docetaxel combination therapy in anthracycline-pretreated patients with advanced breast cancer: phase III trial results. J Clin Oncol. 2002 Jun 15;20(12):2812-23. doi: 10.1200/JCO.2002.09.002. PMID 12065558